CLINICAL TRIAL: NCT01763294
Title: A Controlled Clinical Trial of Cathodal Transcranial Direct Current Stimulation in Patients With Refractory Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez (Other)
Collaborators: Massachusetts General Hospital (Other); University Hospital Freiburg (Other); Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, DANIEL SAN JUAN ORTA, Principal Investigator, El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04/10
Record Dates: First submitted 2013-01-02; First posted 2013-01-08 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Refractory Epilepsy
Keywords: multifocal refractory epilepsy; tDCS; neurostimulation; seizures
MeSH Terms: conditions — Drug Resistant Epilepsy; Seizures | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Nicolet Endeavor CR: 30min (Active Comparator): Apply 1 session of 2 milliampere intensity for 30 minutes. The stimulation mode will be continuous with frequency of 3 Hz. The site of application depends on the basal EEG findings based on the international 10/20 system.
  Interventions: Device: Nicolet Endeavor CR: 30min
- Nicolet Endeavor CR: 60min (Active Comparator): Apply 1 session of 2 milliampere intensity for 60 minutes. The stimulation mode will be continuous with frequency of 3 Hz. The site of application depends on the basal EEG findings based on the international 10/20 system.
  Interventions: Device: Nicolet Endeavor CR: 60min
- Nicolet Endeavor CR: 30min for 3 days (Active Comparator): Apply 3 sessions of 2 milliampere intensity for 30 minutes. The stimulation mode will be continuous with frequency of 3 Hz. The site of application depends on the basal EEG findings based on the international 10/20 system.
  Interventions: Device: Nicolet Endeavor CR: 30min for 3 days
- Nicolet Endeavor CR: 30min for 5 days (Active Comparator): Apply 5 sessions of 2 milliampere intensity for 30 minutes. The stimulation mode will be continuous with frequency of 3 Hz. The site of application depends on the basal EEG findings based on the international 10/20 system.
  Interventions: Device: Nicolet Endeavor CR: 30min for 5 days
- Nicolet Endeavor CR: Placebo (Placebo Comparator): The same procedures just that in this case the machine produces only a 60 second stimulus at the beginning so the patient can feel the initial electric stimulus.
  Interventions: Device: Nicolet Endeavor CR: Placebo

INTERVENTIONS:
Device: Nicolet Endeavor CR: 30min — Transcranial direct current stimulation (tDCS) is a safe, non-invasive method that modulates cortical excitability. In direct current polarization, the cerebral cortex is stimulated through a weak constant electric current in a noninvasive and painless manner. This weak current induces focal changes of cortical excitability increase or decrease depending on the electrode polarity- that last beyond the period of stimulation.
  Other Names: tdcs
  Arms: Nicolet Endeavor CR: 30min
Device: Nicolet Endeavor CR: 60min — Transcranial direct current stimulation (tDCS) is a safe, non-invasive method that modulates cortical excitability. In direct current polarization, the cerebral cortex is stimulated through a weak constant electric current in a noninvasive and painless manner. This weak current induces focal changes of cortical excitability increase or decrease depending on the electrode polarity- that last beyond the period of stimulation.
  Other Names: tdcs
  Arms: Nicolet Endeavor CR: 60min
Device: Nicolet Endeavor CR: 30min for 3 days — Transcranial direct current stimulation (tDCS) is a safe, non-invasive method that modulates cortical excitability. In direct current polarization, the cerebral cortex is stimulated through a weak constant electric current in a noninvasive and painless manner. This weak current induces focal changes of cortical excitability increase or decrease depending on the electrode polarity- that last beyond the period of stimulation.
  Other Names: tdcs
  Arms: Nicolet Endeavor CR: 30min for 3 days
Device: Nicolet Endeavor CR: 30min for 5 days — Transcranial direct current stimulation (tDCS) is a safe, non-invasive method that modulates cortical excitability. In direct current polarization, the cerebral cortex is stimulated through a weak constant electric current in a noninvasive and painless manner. This weak current induces focal changes of cortical excitability increase or decrease depending on the electrode polarity- that last beyond the period of stimulation.
  Other Names: tdcs
  Arms: Nicolet Endeavor CR: 30min for 5 days
Device: Nicolet Endeavor CR: Placebo — The same procedures just that in this case the machine produces only a 60 second stimulus at the beginning so the patient can feel the initial electric stimulus.
  Other Names: placebo
  Arms: Nicolet Endeavor CR: Placebo

SUMMARY:
There is a continuous necessity for the search of new alternatives for safe, affordable and effective noninvasive therapies for patients that are not eligible for focal resective or palliative surgery. The transcranial direct current stimulation (tDCS) therapy has demonstrated to be safe, noninvasive, simple and effective with promising results in case series, case reports and animals models for the treatment of intractable epilepsy. tDCS is a feasible and low cost method to modify cortical excitability in a non-invasive procedure. Its effects on cortical excitability seem to be similar to the effects induced by repetitive transcranial magnetic stimulation. The aim of this study is determine the safety and efficacy in the reduction of the number of seizures (>50%) and epileptiform activity in patients with refractory and multifocal epilepsy after different protocols of tDCS compared with placebo.

DETAILED DESCRIPTION:
This is a prospective interventional clinical study. All enrolled patients have multifocal and refractory epilepsy that voluntarily will accept to participate in the study signing a consent informed form. All patients are from the epilepsy clinic our Institute that meet the criteria. All patients will be randomized and divided in 5 groups (45 patients); placebo group, active group of one session 30 minutes, active group of one session of 60 minutes, active group of 30 minutes for 3 consecutively days and 30 minutes for 5 consecutively days. After the selection, the patients will record their EEG of 30 min in order to register the basal epileptic activity and determine the most epileptic area, where the intervention will be applied. Then, an EEG will be realized after the intervention, one month after and two months after.

The equipment used to apply the therapy is approved for medical use in our country. The equipment is Nicolet, Endeavor used at low amplitude for direct electrical nervous stimulation mode. The intensity to apply will be 2 milliampere. The stimulation mode is continuous with frequency of 3 Hz. The site of application depends on the basal EEG findings, nevertheless, it is ruled by the international EEG 10/20 system.

The cathodal electrode is applies with disposable needle of 12 mm long and 0.5 mm wide, while the anodal electrode is applied with conventional cup electrodes with a 2mm hole in the center an a recording surface of silver chloride /silver. After the intervention the patient is asked about any adverse effect form the therapy application and the EEG is realized as the investigators described before. The patient will receive a follow up dates at one and two months. The patient must make a calendar with the frequency of seizures and must not change the actual medication.

Placebo. This group receives the same procedures just that in this case the machine produces a 60 second stimulus at the beginning so the patient can feel the initial electric stimulus.

The investigators will record the frequency of the seizures and analysis of the epileptiform activity in the EEGs in the baseline, after therapy, 1 month and 2 months of follow-up. As well the safety profile of the tDCS.

ELIGIBILITY:
Inclusion Criteria:

* any gender
* age ≥ 15 and <65 years
* Refractory epilepsy characterized by 3 or more seizures by month and the right use of 2 or more antiepileptic drugs during the last 12 months
* Not eligible for surgery treatment
* Right attachment to the antiepileptic treatment established at least 12 months before the date of inclusion
* Multifocal epilepsy defined as 2 or more lobar regions affected with epileptic activity

Exclusion Criteria:

* Patients with pseudoseizures
* Previous craniotomy
* Active local infection of the skull
* Informed consent not signed
* Patients with generalized idiopathic epilepsy or focal idiopathic epilepsy
* Patients in stupor or coma
* Patients in lactation or pregnancy
* Patients with chronic degenerative diseases of the nervous system
* Patients with exacerbated chronic degenerative diseases

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of seizures | 2 months
  The number of the seizures monthly for 2 months

SECONDARY OUTCOMES:
Frequency of epileptiform discharges | 2 months
  The frequency of the epileptiform discharges on EEGs evaluate at the baseline, after therapy, 1 and 2 months.
Amplitude of epileptiform discharges | 2 monts
  Amplitude of the epileptiform discharges on EEGs evaluate at the baseline, after therapy, 1 and 2 months.

OTHER OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety | 2 months
  Adverse effects reported by the patient during the therapy and the follow-up dates for 1 and 2 months.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel San-juan, MD, Principal Investigator — Instituto Nacional de Neurología y Neurocirugía Manuel Velasco Suárez
Locations (1):
- Instituto Nacional de Neurología y Neurocirugía, Mexico City, Mexico City, Mexico

REFERENCES:
- [Result] San-Juan D, Calcaneo Jde D, Gonzalez-Aragon MF, Bermudez Maldonado L, Avellan AM, Argumosa EV, Fregni F. Transcranial direct current stimulation in adolescent and adult Rasmussen's encephalitis. Epilepsy Behav. 2011 Jan;20(1):126-31. doi: 10.1016/j.yebeh.2010.10.031. Epub 2010 Dec 17. PMID 21167786
- [Result] Fregni F, Thome-Souza S, Nitsche MA, Freedman SD, Valente KD, Pascual-Leone A. A controlled clinical trial of cathodal DC polarization in patients with refractory epilepsy. Epilepsia. 2006 Feb;47(2):335-42. doi: 10.1111/j.1528-1167.2006.00426.x. PMID 16499758
- [Derived] San-Juan D, Espinoza Lopez DA, Vazquez Gregorio R, Trenado C, Fernandez-Gonzalez Aragon M, Morales-Quezada L, Hernandez Ruiz A, Hernandez-Gonzalez F, Alcaraz-Guzman A, Anschel DJ, Fregni F. Transcranial Direct Current Stimulation in Mesial Temporal Lobe Epilepsy and Hippocampal Sclerosis. Brain Stimul. 2017 Jan-Feb;10(1):28-35. doi: 10.1016/j.brs.2016.08.013. Epub 2016 Aug 31. PMID 27693237